CLINICAL TRIAL: NCT00037622
Title: An Open-Label Treatment Protocol to Provide Continued ACH-126,443 to Subjects of Previous Achillion-Sponsored Phase 1 and 2 Studies in Chronic Hepatitis B Infection
Brief Title: Safety and Antiviral Study of ACH-126, 443 (Beta-L-Fd4C) in the Treatment of Adults With Chronic Hepatitis B Infection.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Safety concerns from other studies.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACH443-901
Record Dates: First submitted 2002-05-17; First posted 2002-05-20 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Chronic Hepatitis B
Keywords: E-antigen positive, treatment naïve chronic HBV infected, lamivudine resistant chronic Hepatitis B, Achillion
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — dexelvucitabine

INTERVENTIONS:
Drug: ACH-126, 443 (beta-L-Fd4C)

SUMMARY:
The purpose of this study is to determine the safety and antiviral HBV activity of ACH-126,443 (beta-L-Fd4C) in the treatment of Subjects of Previous Achillion-Sponsored Phase 1 and 2 Studies in Chronic Hepatitis B Infection.

DETAILED DESCRIPTION:
Evaluation of safety and antiviral activity of the 5mg dose of ACH-126,443 for up to three months of treatment in the population described.

ELIGIBILITY:
Inclusion Criteria:

* Participants in previous Phase 1 or 2 trials of ACH-126,443 who met entry criteria for previous studies.
* Adults ? 18 years of age
* Chronic HBV infection, known to be HbsAg positive ? 6 months
* Plasma HBV DNA level ? 100,000 copies/mL prior to initiation of ACH-126,443 in an earlier study
* Plasma HBV DNA level that in the medical judgment of the investigator, warrant's antiviral treatment
* HIV negative
* Basic hematologic and chemistry parameters within acceptable limits (defined in protocol)
* No need for excluded medications
* Subjects of reproductive capability must either practice abstinence or utilize two approved forms of birth control, one of which must be barrier protection (condom with spermicidal, diaphragm with spermicidal)

Exclusion Criteria

* HIV infection
* Active Hepatitis C co-infection
* Concurrent systemic antiviral treatment
* Treatment for HBV infection with lamivudine (3TC) for longer than three (3) months since participation in previous trial of ACH-126,443
* Previous therapy with agents with significant systemic myelosuppressive or cytotoxic potential within 3 months of study start or the expected need for such therapy at study start
* Alcohol abuse
* Pregnancy or breast-feeding
* Inability to tolerate oral medication
* AST>10.0 times the upper limit of normal
* ALT>10.0 times the upper limit of normal
* Any clinical condition or prior therapy that, in the Investigators opinion, would make the subject unsuitable for the study or unable to comply with the dosing requirements
* Use of investigational drug not approved by Medical Monitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Study Completion 2003-05 (Actual)

REFERENCES:
- See also: Related Info — http://www.achillion.com